CLINICAL TRIAL: NCT07069322
Title: The Role of Regional Analgesia in Sleep Quality: Evaluation of Additional Regional Block in Total Abdominal Hysterectomy Patients
Brief Title: The Role of Regional Analgesia in Sleep Quality
Status: Not yet recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emine Yilmaz Guler, Principal Investigator, Haseki Training and Research Hospital
Other Study IDs: TH-220511
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Richards-Campbell Sleep Questionnaire (RCSQ)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Regional: Those who underwent regional analgesic block (GA+RB) in addition to general anesthesia.
  Interventions: Behavioral: Richards-Campbell Sleep Questionnaire (RCSQ)
- Without Regional: Those under general anesthesia (GA)
  Interventions: Behavioral: Richards-Campbell Sleep Questionnaire (RCSQ)

INTERVENTIONS:
Behavioral: Richards-Campbell Sleep Questionnaire (RCSQ) — - Score 0 = Very poor sleep, 100 = Very good sleep

SUMMARY:
To evaluate the effect of regional analgesic blocks (TAP or rectus sheath block) applied in addition to general anesthesia on postoperative sleep quality in patients undergoing total abdominal hysterectomy (RCSQ score).

ELIGIBILITY:
Inclusion Criteria:

* Elective TAH planned
* ASA I-III group
* Female patients aged 18-70 years
* Those who are planned to be hospitalized at least one night in the postoperative period
* Those who have the cognitive capacity to understand and answer the questionnaire

Exclusion Criteria:

* Patients with a history of neurological or psychiatric disease
* Patients diagnosed with sleep disorders
* Patients with sedative/hypnotic drug use
* Patients requiring additional surgical intervention during the operation
* Patients admitted to intensive care unit
* Patients operated with epidural or spinal anesthesia

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women between the ages of 18 and 70 who will undergo TAH operation under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Richards-Campbell Sleep Questionnaire Score (RCSQ) | Postoperative 24 hours
  Clinically ≥50 points: good/moderate sleep quality, <50 points: poor sleep quality

REFERENCES:
- [Result] Ni Eochagain A, Carolan S, Buggy DJ. Regional anaesthesia truncal blocks for acute postoperative pain and recovery: a narrative review. Br J Anaesth. 2024 May;132(5):1133-1145. doi: 10.1016/j.bja.2023.12.020. Epub 2024 Jan 19. PMID 38242803
- [Result] Yang RZ, Li YZ, Liang M, Yu JJ, Chen ML, Qiu JJ, Lin SZ, Wu XD, Zeng K. Stellate Ganglion Block Improves Postoperative Sleep Quality and Analgesia in Patients with Breast Cancer: A Randomized Controlled Trial. Pain Ther. 2023 Apr;12(2):491-503. doi: 10.1007/s40122-022-00473-y. Epub 2023 Jan 18. PMID 36652140